CLINICAL TRIAL: NCT03205371
Title: Immunogenicity and Safety of an Investigational Quadrivalent Meningococcal Conjugate Vaccine Administered Concomitantly With Other Pediatric Vaccines in Healthy Toddlers
Brief Title: Immunogenicity and Safety of a Meningococcal Conjugate Vaccine Given Concomitantly With Other Vaccines in Toddlers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MET57; U1111-1161-2787 (Other: WHO Universal Trial Number (UTN))
Record Dates: First submitted 2017-06-28; First posted 2017-07-02 (Actual); Results first posted 2020-06-09 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Meningitis, Meningococcal
Keywords: Meningitis; Meningococcal Meningitis; Meningococcal Infections; MenACYW Conjugate vaccine
MeSH Terms: conditions — Meningitis, Meningococcal; Meningitis; Meningococcal Infections

STUDY DESIGN:
Intervention Model Description: Phase III, open-label, randomized, parallel-group, active-controlled, multicenter study
Who Masked: Outcomes Assessor
Masking Description: The study had an open-label design; however, as per the protocol, the laboratory technicians who were responsible for performing the serological testing remained blinded to the participants' group allocations throughout the study to avoid any bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (12):
- South Korea(Group1):MenACYW Conjugate + MMR+ Varicella Vaccine (Experimental): Healthy, meningococcal-vaccine naïve toddlers (aged 12 to 23 months) received single dose of MenACYW Conjugate vaccine, MMR vaccine, and varicella vaccine on Day 0.
  Interventions: Biological: MenACYW conjugate vaccine; Biological: MMR; Biological: Varicella
- South Korea (Group 2): MenACYW Conjugate Vaccine (Experimental): Healthy, meningococcal-vaccine naïve toddlers (aged 12 to 23 months) received single dose of MenACYW Conjugate vaccine on Day 0.
  Interventions: Biological: MenACYW conjugate vaccine
- South Korea (Group 3): MMR + Varicella Vaccine (Active Comparator): Healthy, meningococcal-vaccine naïve toddlers (aged 12 to 23 months) received single dose of MMR vaccine and varicella vaccine on Day 0.
  Interventions: Biological: MMR; Biological: Varicella
- Thailand (Group 10):MenACYW Conjugate +MMR+Varicella Vaccine (Experimental): Healthy, meningococcal-vaccine naïve toddlers (aged 12 to 23 months) received single dose of MenACYW Conjugate vaccine, MMR vaccine, and varicella vaccine on Day 0.
  Interventions: Biological: MenACYW conjugate vaccine; Biological: MMR; Biological: Varicella
- Thailand (Group 11):MenACYW Conjugate Vaccine (Experimental): Healthy, meningococcal-vaccine naïve toddlers (aged 12 to 23 months) received single dose of MenACYW Conjugate vaccine on Day 0.
  Interventions: Biological: MenACYW conjugate vaccine
- Thailand (Group 12): MMR + Varicella Vaccine (Active Comparator): Healthy, meningococcal-vaccine naïve toddlers (aged 12 to 23 months) received single dose of MMR vaccine and varicella vaccine on Day 0.
  Interventions: Biological: MMR; Biological: Varicella
- Mexico (Group 4): MenACYW Conjugate + DTaP-IPV-HB-Hib Vaccine (Experimental): Healthy, meningococcal-vaccine naïve toddlers (aged 12 to 23 months) received single dose of MenACYW Conjugate vaccine and diphtheria, tetanus, acellular pertussis, hepatitis B, poliomyelitis and Haemophilus influenzae type-b (DTaP-IPV-HB-Hib) vaccine on Day 0.
  Interventions: Biological: MenACYW conjugate vaccine; Biological: DTaP-IPV-HB-Hib
- Mexico (Group 5): MenACYW Conjugate Vaccine (Experimental): Healthy, meningococcal-vaccine naïve toddlers (aged 12 to 23 months) received single dose of MenACYW Conjugate vaccine on Day 0.
  Interventions: Biological: MenACYW conjugate vaccine
- Mexico (Group 6): DTaP-IPV-HB-Hib Vaccine (Active Comparator): Healthy, meningococcal-vaccine naïve toddlers (aged 12 to 23 months) received single dose of DTaP-IPV-HB-Hib vaccine on Day 0.
  Interventions: Biological: DTaP-IPV-HB-Hib
- Russian Federation (Group7): MenACYW Conjugate + PCV13 Vaccine (Experimental): Healthy, meningococcal-vaccine naïve toddlers (aged 15 to 23 months) received single dose of MenACYW Conjugate vaccine and pneumococcal Conjugate vaccine (PCV13) on Day 0.
  Interventions: Biological: MenACYW conjugate vaccine; Biological: PCV13
- Russian Federation (Group 8): MenACYW Conjugate Vaccine (Experimental): Healthy, meningococcal-vaccine naïve toddlers (aged 12 to 14 months or 16 to 23 months) received single dose of MenACYW Conjugate vaccine on Day 0.
  Interventions: Biological: MenACYW conjugate vaccine
- Russian Federation (Group 9): PCV13 Vaccine (Active Comparator): Healthy, meningococcal-vaccine naïve toddlers (aged 15 to 23 months) received single dose of PCV13 vaccine on Day 0.
  Interventions: Biological: PCV13

INTERVENTIONS:
Biological: MenACYW conjugate vaccine — Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus Toxoid Conjugate Vaccine; 0.5 milliliter (mL), Intramuscular
  Arms: Mexico (Group 4): MenACYW Conjugate + DTaP-IPV-HB-Hib Vaccine; Mexico (Group 5): MenACYW Conjugate Vaccine; Russian Federation (Group 8): MenACYW Conjugate Vaccine; Russian Federation (Group7): MenACYW Conjugate + PCV13 Vaccine; South Korea (Group 2): MenACYW Conjugate Vaccine; South Korea(Group1):MenACYW Conjugate + MMR+ Varicella Vaccine; Thailand (Group 10):MenACYW Conjugate +MMR+Varicella Vaccine; Thailand (Group 11):MenACYW Conjugate Vaccine
Biological: MMR — Measles, Mumps, and Rubella Virus Vaccine Live; 0.5 mL, Subcutaneous
  Arms: South Korea (Group 3): MMR + Varicella Vaccine; South Korea(Group1):MenACYW Conjugate + MMR+ Varicella Vaccine; Thailand (Group 10):MenACYW Conjugate +MMR+Varicella Vaccine; Thailand (Group 12): MMR + Varicella Vaccine
Biological: Varicella — Varicella Virus Vaccine Live; 0.5 mL, Subcutaneous
  Arms: South Korea (Group 3): MMR + Varicella Vaccine; South Korea(Group1):MenACYW Conjugate + MMR+ Varicella Vaccine; Thailand (Group 10):MenACYW Conjugate +MMR+Varicella Vaccine; Thailand (Group 12): MMR + Varicella Vaccine
Biological: DTaP-IPV-HB-Hib — Diphtheria, Tetanus, Pertussis (acellular component), Hepatitis B, Poliomyelitis (inactivated), and Haemophilus influenzae type-b conjugate vaccine (adsorbed); 0.5 mL, Intramuscular
  Arms: Mexico (Group 4): MenACYW Conjugate + DTaP-IPV-HB-Hib Vaccine; Mexico (Group 6): DTaP-IPV-HB-Hib Vaccine
Biological: PCV13 — Pneumococcal 13-valent Conjugate Vaccine; 0.5 mL, Intramuscular
  Arms: Russian Federation (Group 9): PCV13 Vaccine; Russian Federation (Group7): MenACYW Conjugate + PCV13 Vaccine

SUMMARY:
This Phase III, open-label, randomized, parallel-group, active-controlled, multicenter study was conducted to assess the immunogenicity and safety of a single dose of Meningococcal Polysaccharide (Serogroups A, C, Y and W) Tetanus Toxoid (MenACYW) Conjugate vaccine when administered alone and in combination with other pediatric vaccines in healthy toddlers in South Korea, Thailand, the Russian Federation, and Mexico.

Primary Objective:

* To describe the immunogenicity profile of MenACYW Conjugate vaccine administered alone or concomitantly with licensed pediatric vaccine(s) (measles-mumps-rubella vaccine [MMR] + Varicella, diphtheria, tetanus, acellular pertussis, hepatitis B, poliomyelitis, and Haemophilus influenzae type-b Conjugate vaccine [DTaP-IPV-HB-Hib], or pneumococcal Conjugate vaccine [PCV13]).

Secondary Objective:

* To describe the immunogenicity profile of licensed pediatric vaccine(s) (MMR + Varicella, DTaP-IPV-HB-Hib, or PCV13) when administered alone or concomitantly with MenACYW Conjugate vaccine.

DETAILED DESCRIPTION:
Healthy, meningococcal-vaccine naïve toddlers aged 12 to 23 months were randomized either to a single dose of MenACYW Conjugate vaccine alone or in combination with other pediatric vaccines in healthy toddlers in South Korea and Thailand (MMR + varicella vaccine), the Russian Federation (PCV13), and Mexico (DTaP-IPV-HB-Hib). Immunogenicity (pre- and 30 days post-vaccination) and safety was assessed.

ELIGIBILITY:
Inclusion Criteria:

* For South Korea: Korean males and females aged 12 to 23 months on the day of the first study visit.
* For Mexico: Males and females aged 12 to 23 months on the day of the first study visit.
* For the Russian Federation: Males and females aged 12 to 14 months or 16 to 23 months on the day of the first study visit (eligible for enrollment to MenACYW Conjugate vaccine group) or 15 to 23 months on the day of the first study visit (eligible for enrollment to the MenACYW Conjugate vaccine positive(+) PCV13 group or the PCV13 group).
* For Thailand: Thai males and females aged 12 to 23 months on the day of the first study visit
* Participants had received all recommended standard of care vaccinations according to their age as per local regulations*.
* For the Russian Federation only, participants aged 15 to 23 months on the day of the first study visit (eligible for enrollment to MenACYW Conjugate vaccine+PCV13 group or the PCV13 group) must not had received the third PCV13 vaccination corresponding to his or her age as per the country's National Immunization Program (NIP). The 2nd dose of PCV13 must had been administered at least 4 weeks before the 3rd dose of PCV13 was administered in the study.
* For South Korea, participants must not had received the MMR or Varicella vaccination corresponding to his or her age at inclusion.
* For Mexico, participants must not had received the DTaP-IPV-HB-Hib vaccination corresponding to his or her age at inclusion.
* For Thailand, participants must not have received the any dose of MMR or V vaccination.
* Informed consent form was signed and dated by the parent(s) or guardian if allowed by local regulations (and by independent witnesses if required by local regulations)†.
* Participant and parent/guardian were able to attend all scheduled visits and to comply with all trial procedures.
* *Participants must had received the total number of doses expected for each vaccine recommended for his/her age in the respective NIPs, but inclusion of participants with variations in the vaccine administration timeframes is considered acceptable if the total number of doses for the corresponding vaccines had been completed (e.g., in Mexico, 3 infant doses of the pentavalent vaccine must had been administered but the 4th dose due in the 2nd year of life should not had been administered for participants to be included in the trial). For the Russian Federation only, participants that had not received a seasonal flu vaccination from 6 months of age according to the Russian NIP were still eligible to participate in this study. For Thailand only, participants who had received a vaccine ahead of the schedule can still be included in the study provided the first doses of MMR and Varicella vaccines have not been administered prior to inclusion.
* †In the Russian Federation, as per local regulations, only the participant's parent(s) are entitled to sign an informed consent form. A child under the responsibility of a guardian were not included in the study.

Exclusion Criteria:

* Participation in the 4 weeks preceding the first trial vaccination or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure.
* Receipt of any vaccine in the 4 weeks (28 days) preceding the first trial vaccination or planned receipt of any vaccine prior to Visit 2 except for influenza vaccination, which may be received at least 2 weeks before or after the study investigational vaccines. This exception includes monovalent pandemic influenza vaccines and multivalent influenza vaccines.
* Previous vaccination against meningococcal disease with either the trial vaccine or another vaccine (i.e., mono- or polyvalent, polysaccharide, or conjugate meningococcal vaccine containing serogroups A, C, Y, or W; or meningococcal B vaccine).
* For participants enrolled at sites in the Russian Federation: previous vaccination with the third dose of PCV13 in participants 15 to 23 months of age (eligible for MenACYW Conjugate vaccine+PCV13 group or the PCV13).
* For participants enrolled at sites in Mexico: known history of seizures, or uncontrolled neurologic disorder (including epilepsy); or encephalopathy of unknown etiology occurring within 7 days following previous vaccination with pertussis containing vaccine; previous vaccination with DTaP-IPV-HB-Hib or DTaP-containing vaccine at 12 to 23 months of age.
* For participants enrolled at sites in South Korea and Thailand: known history of seizures, cerebral injury, or encephalopathy; previous vaccination with MMR or Varicella at 12 to 23 months of age.
* Receipt of immune globulins, blood or blood-derived products in the past 3 months.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* History of meningococcal infection, confirmed either clinically, serologically, or microbiologically.
* At high risk for meningococcal infection during the trial, according to the Investigator's judgment (specifically, but not limited to, participants with persistent complement deficiency, with anatomic or functional asplenia, or participants traveling to countries with high endemic or epidemic disease).
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine(s) used in the trial or to a vaccine containing any of the same substances.
* Verbal report of thrombocytopenia, as reported by the parent/guardian, contraindicating intramuscular (IM) vaccination by the Investigator's judgment.
* Known bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM vaccination by the Investigator's judgment.
* Personal history of Guillain-Barré syndrome (GBS).
* Personal history of an Arthus-like reaction after vaccination with a tetanus toxoid-containing vaccine.
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion.
* For participants enrolled at sites in South Korea or Mexico and Thailand: Moderate or severe acute illness/infection (according to investigator's judgment) on the day of vaccination or febrile illness (temperature >= 38.0 degree Celsius [°C]). A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided.
* For participants enrolled at sites in the Russian Federation: Acute disease of any severity on the day of vaccination or febrile illness (axillary temperature >= 37.0°C). A prospective participant should not be included in the study until the condition has resolved or the febrile event had subsided.
* Receipt of oral or injectable antibiotic therapy within 72 hours prior to the first blood draw.
* Identified as a natural or adopted child of the Investigator or employee with direct involvement in the proposed study.

Ages: 12 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1183 (Actual)
Dates: Start 2016-11-07 (Actual); Primary Completion 2018-07-19 (Actual); Study Completion 2018-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (29):
- Mexico (3):
  - Acapulco
  - Mexico City
  - Tlaltizapán
- Russia (12):
  - Barnaul
  - Kazan'
  - Krasnodar
  - Moscow
  - Murmansk
  - Novosibirsk
  - Perm
  - Saint Petersburg
  - Samara
  - Smolensk
  - Tomsk
  - Yekaterinburg
- South Korea (12):
  - Ansan
  - Anyang
  - Daegu
  - Daejeon
  - Gwangju
  - Ilsan
  - Incheon
  - Jeju City
  - Seoul
  - Suwon
  - Wŏnju
  - Yangsan
- Thailand (2):
  - Pathum Wan, Bangkok
  - Rajthevi, Bangkok

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Dhingra MS, Namazova-Baranova L, Arredondo-Garcia JL, Kim KH, Limkittikul K, Jantarabenjakul W, Perminova O, Kobashi IAR, Bae CW, Ojeda J, Park J, Chansinghakul D, B'Chir S, Neveu D, Bonaparte M, Jordanov E. Immunogenicity and safety of a quadrivalent meningococcal tetanus toxoid-conjugate vaccine administered concomitantly with other paediatric vaccines in toddlers: a phase III randomised study. Epidemiol Infect. 2021 Apr 5;149:e90. doi: 10.1017/S0950268821000698. PMID 33814028
- See also: Related info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled in South Korea, Mexico, the Russian Federation, and Thailand from 07 November 2016 to 13 June 2018.
Pre-assignment Details: A total of 1183 participants were enrolled and randomized in the study.
Groups:
- South Korea(Group1):MenACYW Conjugate +MMR +Varicella Vaccine: Healthy, meningococcal-vaccine naïve toddlers (aged 12 to 23 months) received single dose of Meningococcal Polysaccharide (Serogroups A, C, Y and W) Tetanus Toxoid (MenACYW) Conjugate vaccine, measles-mumps-rubella (MMR) vaccine, and varicella vaccine on Day 0.
- Thailand (Group 10):MenACYW Conjugate + MMR+ Varicella Vaccine: Healthy, meningococcal-vaccine naïve toddlers (aged 12 to 23 months) received single dose of MenACYW Conjugate vaccine, MMR vaccine, and varicella vaccine on Day 0.
- Thailand (Group 11): MenACYW Conjugate Vaccine; Mexico (Group 5): MenACYW Conjugate Vaccine: Healthy, meningococcal-vaccine naïve toddlers (aged 12 to 23 months) received single dose of MenACYW Conjugate vaccine on Day 0.
- Russian Federation (Group7): MenACYW Conjugate + PCV13 Vaccine: Healthy, meningococcal-vaccine naïve toddlers (aged 15 to 23 months) received single dose of MenACYW Conjugate and pneumococcal Conjugate vaccine (PCV13) on Day 0.
Period: Overall Study
Arm/Group | South Korea(Group1):MenACYW Conjugate +MMR +Varicella Vaccine | South Korea (Group 2): MenACYW Conjugate Vaccine | South Korea (Group 3): MMR + Varicella Vaccine | Thailand (Group 10):MenACYW Conjugate + MMR+ Varicella Vaccine | Thailand (Group 11): MenACYW Conjugate Vaccine | Thailand (Group 12): MMR + Varicella Vaccine | Mexico (Group 4): MenACYW Conjugate + DTaP-IPV-HB-Hib Vaccine | Mexico (Group 5): MenACYW Conjugate Vaccine | Mexico (Group 6): DTaP-IPV-HB-Hib Vaccine | Russian Federation (Group7): MenACYW Conjugate + PCV13 Vaccine | Russian Federation (Group 8): MenACYW Conjugate Vaccine | Russian Federation (Group 9): PCV13 Vaccine
Started | 107 | 53 | 53 | 86 | 42 | 42 | 200 | 100 | 100 | 200 | 100 | 100
Safety Analysis Set (SafAS) (SafAS: participants who received at least 1 dose of study vaccine(s) & had any safety data available) | 103 | 52 | 53 | 86 | 42 | 42 | 200 | 100 | 100 | 200 | 100 | 99
Per-protocol Analysis Set (PPAS) (PPAS: participants who received at least 1 dose of study vaccine, and had no protocol deviations.) | 92 | 45 | 50 | 85 | 42 | 42 | 155 | 79 | 68 | 196 | 96 | 92
Completed | 103 | 52 | 53 | 86 | 42 | 42 | 190 | 97 | 95 | 200 | 100 | 99
Not Completed | 4 | 1 | 0 | 0 | 0 | 0 | 10 | 3 | 5 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 4 | 1 | 0 | 0 | 0 | 0 | 4 | 0 | 2 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 2 | 3 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants.
Groups:
- South Korea(Group1):MenACYW Conjugate +MMR+ Varicella Vaccine; Thailand (Group 10): MenACYW Conjugate + MMR+Varicella Vaccine: Healthy, meningococcal-vaccine naïve toddlers (aged 12 to 23 months) received single dose of MenACYW Conjugate vaccine, MMR vaccine, and varicella vaccine on Day 0.
- Mexico (Group 4): MenACYW Conjugate + DTaP-IPV-HB-Hib Vaccine: Healthy, meningococcal-vaccine naïve toddlers (aged 12 to 23 months) received single dose of MenACYW Conjugate vaccine and DTaP-IPV-HB-Hib vaccine on Day 0.
- Total: Total of all reporting groups
Arm/Group | South Korea(Group1):MenACYW Conjugate +MMR+ Varicella Vaccine | South Korea (Group 2): MenACYW Conjugate Vaccine | South Korea (Group 3): MMR + Varicella Vaccine | Thailand (Group 10): MenACYW Conjugate + MMR+Varicella Vaccine | Thailand (Group 11): MenACYW Conjugate Vaccine | Thailand (Group 12): MMR + Varicella Vaccine | Mexico (Group 4): MenACYW Conjugate + DTaP-IPV-HB-Hib Vaccine | Mexico (Group 5): MenACYW Conjugate Vaccine | Mexico (Group 6): DTaP-IPV-HB-Hib Vaccine | Russian Federation (Group7): MenACYW Conjugate + PCV13 Vaccine | Russian Federation (Group 8): MenACYW Conjugate Vaccine | Russian Federation (Group 9): PCV13 Vaccine | Total
Number analyzed (Participants) | 107 | 53 | 53 | 86 | 42 | 42 | 200 | 100 | 100 | 200 | 100 | 100 | 1183
Age, Continuous [Mean (Standard Deviation); unit: months] | 12.7 (1.58) | 12.7 (1.50) | 12.3 (0.96) | 12.4 (0.90) | 12.4 (0.88) | 12.8 (1.76) | 16.4 (2.73) | 16.8 (2.83) | 16.8 (2.99) | 16.5 (2.36) | 16.0 (3.10) | 16.3 (2.26) | 15.2 (2.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 18 | 29 | 47 | 23 | 23 | 93 | 46 | 48 | 78 | 51 | 45 | 550
  Male | 58 | 35 | 24 | 39 | 19 | 19 | 107 | 54 | 52 | 122 | 49 | 55 | 633
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 86 | 42 | 42 | 0 | 0 | 1 | 2 | 1 | 4 | 179
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0 | 200 | 100 | 99 | 198 | 99 | 96 | 792
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 106 | 53 | 53 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 212
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 107 | 53 | 53 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 213
  Mexico | 0 | 0 | 0 | 0 | 0 | 0 | 200 | 100 | 100 | 0 | 0 | 0 | 400
  Russia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 200 | 100 | 100 | 400
  Thailand | 0 | 0 | 0 | 86 | 42 | 42 | 0 | 0 | 0 | 0 | 0 | 0 | 170

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers of Meningococcal Serogroups A, C, Y, and W Antibodies Following Injection With MenACYW Conjugate Vaccine Administered Alone or Concomitantly With Other Pediatric Vaccines: Groups 1, 2, 4, 5, 7, 8, 10, and 11
Description: Antibody titers of Meningococcal Serogroups A, C, Y, and W were measured by serum bactericidal assay using human complement (hSBA) assay. Data for this outcome measure was planned to reported for the combined population of Groups 1 and 10, Groups 2 and 11.
Time Frame: Day 0 and Day 30 post-vaccination
Population: Analysis was performed on PPAS which included participants who received at least one dose of the study vaccine(s), had a valid post-vaccination blood sample result and no protocol deviations. Data for this outcome measure were not planned to be collected and analyzed for Groups 3, 6, 9, and 12.
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Groups:
- Groups 1and10: MenACYW Conjugate Vaccine+MMR+Varicella Vaccine: Healthy, meningococcal-vaccine naïve toddlers (aged 12 to 23 months) from South Korea and Thailand received single dose of MenACYW Conjugate vaccine, MMR vaccine, and varicella vaccine on Day 0.
- Groups 2 and 11: MenACYW Conjugate Vaccine: Healthy, meningococcal-vaccine naïve toddlers (aged 12 to 23 months) from South Korea and Thailand received single dose of MenACYW Conjugate vaccine on Day 0.
- Russian Federation (Group 7): MenACYW Conjugate +PCV13 Vaccine: Healthy, meningococcal-vaccine naïve toddlers (aged 15 to 23 months) received single dose of MenACYW Conjugate vaccine and PCV13 vaccine on Day 0.
Arm/Group | Groups 1and10: MenACYW Conjugate Vaccine+MMR+Varicella Vaccine | Groups 2 and 11: MenACYW Conjugate Vaccine | Mexico (Group 4): MenACYW Conjugate + DTaP-IPV-HB-Hib Vaccine | Mexico (Group 5): MenACYW Conjugate Vaccine | Russian Federation (Group 7): MenACYW Conjugate +PCV13 Vaccine | Russian Federation (Group 8): MenACYW Conjugate Vaccine
Number analyzed (Participants) | 177 | 87 | 155 | 79 | 196 | 96
titers (1/dilution)
  Serogroup A: Day 0 | 5.20 [4.56 to 5.93] | 6.10 [5.00 to 7.44] | 5.35 [4.82 to 5.94] | 5.49 [4.66 to 6.45] | 5.99 [5.30 to 6.76] | 8.54 [6.47 to 11.3]
  Serogroup A: Day 30 | 43.9 [37.4 to 51.6] | 30.0 [23.1 to 39.0] | 31.4 [25.9 to 38.1] | 37.8 [28.5 to 50.2] | 24.6 [20.2 to 30.1] | 49.0 [36.8 to 65.3]
  Serogroup C: Day 0 | 2.37 [2.11 to 2.65] | 2.58 [2.15 to 3.10] | 2.21 [2.11 to 2.31] | 2.16 [2.00 to 2.34] | 2.77 [2.43 to 3.16] | 3.69 [2.84 to 4.81]
  Serogroup C: Day 30 | 876 [725 to 1057] | 600 [456 to 790] | 749 [633 to 886] | 666 [538 to 825] | 205 [156 to 269] | 309 [218 to 437]
  Serogroup Y: Day 0 | 3.14 [2.78 to 3.54] | 3.12 [2.58 to 3.78] | 2.63 [2.37 to 2.92] | 2.94 [2.45 to 3.53] | 2.90 [2.56 to 3.28] | 3.49 [2.68 to 4.53]
  Serogroup Y: Day 30 | 88.9 [75.1 to 105] | 60.0 [47.3 to 76.3] | 79.7 [65.7 to 96.6] | 90.9 [66.8 to 124] | 139 [111 to 173] | 172 [130 to 229]
  Serogroup W: Day 0 | 2.15 [2.00 to 2.30] | 2.31 [2.02 to 2.64] | 2.41 [2.22 to 2.62] | 2.16 [2.04 to 2.30] | 2.93 [2.54 to 3.38] | 3.62 [2.73 to 4.79]
  Serogroup W: Day 30 | 46.8 [39.1 to 56.0] | 35.5 [27.6 to 45.7] | 40.0 [32.5 to 49.3] | 50.9 [37.2 to 69.8] | 57.4 [47.9 to 68.6] | 57.0 [44.3 to 73.5]

2. Primary Outcome: Percentage of Participants With Antibody Titers >=1:4 and >=1:8 Against Meningococcal Serogroups A, C, Y, and W Following Injection With MenACYW Conjugate Vaccine Administered Alone or With Other Pediatric Vaccines: Groups 1, 2, 4, 5, 7, 8, 10, and 11
Description: Antibody titers of Meningococcal Serogroups A, C, Y, and W were measured by hSBA assay. Data for this outcome measure was planned to be reported for the combined population of Groups 1 and 10, Groups 2 and 11.
Time Frame: Day 0 and Day 30 post-vaccination
Population: Analysis was performed on PPAS. Data for this outcome measure were not planned to be collected and analyzed for Groups 3, 6, 9, and 12.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Groups 1and 10:MenACYW Conjugate Vaccine+MMR+Varicella Vaccine: Healthy, meningococcal-vaccine naïve toddlers (aged 12 to 23 months) from South Korea and Thailand received single dose of MenACYW Conjugate vaccine, MMR vaccine, and varicella vaccine on Day 0.
Arm/Group | Groups 1and 10:MenACYW Conjugate Vaccine+MMR+Varicella Vaccine | Groups 2 and 11: MenACYW Conjugate Vaccine | Mexico (Group 4): MenACYW Conjugate + DTaP-IPV-HB-Hib Vaccine | Mexico (Group 5): MenACYW Conjugate Vaccine | Russian Federation (Group 7): MenACYW Conjugate +PCV13 Vaccine | Russian Federation (Group 8): MenACYW Conjugate Vaccine
Number analyzed (Participants) | 177 | 87 | 155 | 79 | 196 | 96
percentage of participants
  Serogroup A: Day 0 (>=1:4) | 75.1 [68.1 to 81.3] | 82.8 [73.2 to 90.0] | 82.6 [75.7 to 88.2] | 82.3 [72.1 to 90.0] | 82.1 [76.1 to 87.2] | 85.4 [76.7 to 91.8]
  Serogroup A: Day 0 (>=1:8) | 37.9 [30.7 to 45.4] | 44.8 [34.1 to 55.9] | 45.8 [37.8 to 54.0] | 46.8 [35.5 to 58.4] | 49.0 [41.8 to 56.2] | 54.2 [43.7 to 64.4]
  Serogroup A: Day 30 (>=1:4) | 98.9 [96.0 to 99.9] | 95.4 [88.6 to 98.7] | 98.1 [94.4 to 99.6] | 97.5 [91.2 to 99.7] | 94.9 [90.8 to 97.5] | 97.9 [92.7 to 99.7]
  Serogroup A: Day 30 (>=1:8) | 97.7 [94.3 to 99.4] | 92.0 [84.1 to 96.7] | 92.9 [87.7 to 96.4] | 89.9 [81.0 to 95.5] | 83.7 [77.7 to 88.6] | 90.6 [82.9 to 95.6]
  Serogroup C: Day 0 (>=1:4) | 9.6 [5.7 to 14.9] | 16.1 [9.1 to 25.5] | 12.3 [7.5 to 18.5] | 7.6 [2.8 to 15.8] | 19.9 [14.5 to 26.2] | 36.5 [26.9 to 46.9]
  Serogroup C: Day 0 (>=1:8) | 4.0 [1.6 to 8.0] | 6.9 [2.6 to 14.4] | 1.9 [0.4 to 5.6] | 1.3 [0.0 to 6.9] | 8.7 [5.1 to 13.5] | 17.7 [10.7 to 26.8]
  Serogroup C: Day 30 (>=1:4) | 100.0 [97.9 to 100.0] | 100.0 [95.8 to 100.0] | 100.0 [97.6 to 100.0] | 100.0 [95.4 to 100.0] | 98.5 [95.6 to 99.7] | 99.0 [94.3 to 100.0]
  Serogroup C: Day 30 (>=1:8) | 100.0 [97.9 to 100.0] | 100.0 [95.8 to 100.0] | 100.0 [97.6 to 100.0] | 100.0 [95.4 to 100.0] | 93.9 [89.5 to 96.8] | 99.0 [94.3 to 100.0]
  Serogroup Y: Day 0 (>=1:4) | 32.2 [25.4 to 39.6] | 28.7 [19.5 to 39.4] | 19.4 [13.5 to 26.5] | 25.3 [16.2 to 36.4] | 21.9 [16.4 to 28.4] | 32.3 [23.1 to 42.6]
  Serogroup Y: Day 0 (>=1:8) | 18.6 [13.2 to 25.2] | 17.2 [10.0 to 26.8] | 11.0 [6.5 to 17.0] | 12.7 [6.2 to 22.0] | 14.3 [9.7 to 20.0] | 15.6 [9.0 to 24.5]
  Serogroup Y: Day 30 (>=1:4) | 99.4 [96.9 to 100.0] | 96.6 [90.3 to 99.3] | 98.7 [95.4 to 99.8] | 100.0 [95.4 to 100.0] | 98.5 [95.6 to 99.7] | 99.0 [94.3 to 100.0]
  Serogroup Y: Day 30 (>=1:8) | 99.4 [96.9 to 100.0] | 95.4 [88.6 to 98.7] | 98.7 [95.4 to 99.8] | 98.7 [93.1 to 100.0] | 97.4 [94.1 to 99.2] | 97.9 [92.7 to 99.7]
  Serogroup W: Day 0 (>=1:4) | 5.1 [2.4 to 9.4] | 11.5 [5.7 to 20.1] | 14.8 [9.6 to 21.4] | 8.9 [3.6 to 17.4] | 16.8 [11.9 to 22.8] | 26.0 [17.6 to 36.0]
  Serogroup W: Day 0 (>=1:8) | 1.1 [0.1 to 4.0] | 2.3 [0.3 to 8.1] | 7.7 [4.1 to 13.1] | 2.5 [0.3 to 8.8] | 12.8 [8.4 to 18.3] | 20.8 [13.2 to 30.3]
  Serogroup W: Day 30 (>=1:4) | 98.9 [96.0 to 99.9] | 96.6 [90.3 to 99.3] | 97.4 [93.5 to 99.3] | 96.2 [89.3 to 99.2] | 95.9 [92.1 to 98.2] | 96.9 [91.1 to 99.4]
  Serogroup W: Day 30 (>=1:8) | 96.0 [92.0 to 98.4] | 92.0 [84.1 to 96.7] | 90.3 [84.5 to 94.5] | 92.4 [84.2 to 97.2] | 94.4 [90.2 to 97.2] | 95.8 [89.7 to 98.9]

3. Primary Outcome: Percentage of Participants With >=4-Fold Rise in Antibody Titers Against Meningococcal Serogroups A, C, Y, and W Following Injection With MenACYW Conjugate Vaccine Administered Alone or With Other Pediatric Vaccines: Groups 1, 2, 4, 5, 7, 8, 10, and 11
Description: as for outcome 2
Time Frame: Day 0 up to Day 30 post-vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Groups 1 and10:MenACYW Conjugate Vaccine+MMR+Varicella Vaccine: Healthy, meningococcal-vaccine naïve toddlers (aged 12 to 23 months) from South Korea and Thailand received single dose of MenACYW Conjugate vaccine, MMR vaccine, and varicella vaccine on Day 0.
- Russian Federation (Group 7): MenACYW Conjugate +PCV13 Vaccine: Healthy, meningococcal-vaccine naïve toddlers (aged 15 to 23 months) received single dose of MenACYW Conjugate and PCV13 vaccine on Day 0.
Arm/Group | Groups 1 and10:MenACYW Conjugate Vaccine+MMR+Varicella Vaccine | Groups 2 and 11: MenACYW Conjugate Vaccine | Mexico (Group 4): MenACYW Conjugate + DTaP-IPV-HB-Hib Vaccine | Mexico (Group 5): MenACYW Conjugate Vaccine | Russian Federation (Group 7): MenACYW Conjugate +PCV13 Vaccine | Russian Federation (Group 8): MenACYW Conjugate Vaccine
Number analyzed (Participants) | 177 | 87 | 155 | 79 | 196 | 96
percentage of participants
  Serogroup A | 82.5 [76.1 to 87.8] | 64.4 [53.4 to 74.4] | 69.0 [61.1 to 76.2] | 70.9 [59.6 to 80.6] | 58.2 [50.9 to 65.2] | 72.9 [62.9 to 81.5]
  Serogroup C | 98.3 [95.1 to 99.6] | 98.9 [93.8 to 100.0] | 100.0 [97.6 to 100.0] | 98.7 [93.1 to 100.0] | 92.3 [87.7 to 95.7] | 91.7 [84.2 to 96.3]
  Serogroup Y | 95.5 [91.3 to 98.0] | 89.7 [81.3 to 95.2] | 96.8 [92.6 to 98.9] | 94.9 [87.5 to 98.6] | 94.4 [90.2 to 97.2] | 93.8 [86.9 to 97.7]
  Serogroup W | 94.9 [90.6 to 97.6] | 89.7 [81.3 to 95.2] | 86.5 [80.0 to 91.4] | 92.4 [84.2 to 97.2] | 88.8 [83.5 to 92.8] | 90.6 [82.9 to 95.6]

4. Primary Outcome: Percentage of Participants Achieving hSBA Vaccine Seroresponse for Meningococcal Serogroups A, C, Y, and W Following Injection With MenACYW Conjugate Vaccine Administered Alone or Concomitantly With Pediatric Vaccines: Groups 1, 2, 4, 5, 7, 8, 10, and 11
Description: The hSBA vaccine seroresponse for serogroups A, C, Y, and W was defined as post-vaccination hSBA titers >=1:16 for participants with pre-vaccination titers <1:8 or at least a 4-fold increase in post-vaccination hSBA titers from pre- to post-vaccination, for participants with pre-vaccination titers >=1:8. Data for this outcome measure was planned to be reported for the combined population of Groups 1 and 10, Groups 2 and 11.
Time Frame: Day 30 post-vaccination
Population: Analysis was performed on PPAS. Data for this outcome measure were not planned to be collected and analyzed for Groups 3, 6, 9 and 12.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Groups 1 and10:MenACYW Conjugate Vaccine+MMR+Varicella Vaccine | Groups 2 and 11: MenACYW Conjugate Vaccine | Mexico (Group 4): MenACYW Conjugate + DTaP-IPV-HB-Hib Vaccine | Mexico (Group 5): MenACYW Conjugate Vaccine | Russian Federation (Group 7): MenACYW Conjugate +PCV13 Vaccine | Russian Federation (Group 8): MenACYW Conjugate Vaccine
Number analyzed (Participants) | 177 | 87 | 155 | 79 | 196 | 96
percentage of participants
  Serogroup A | 78.5 [71.7 to 84.3] | 63.2 [52.2 to 73.3] | 67.1 [59.1 to 74.4] | 69.6 [58.2 to 79.5] | 56.1 [48.9 to 63.2] | 71.9 [61.8 to 80.6]
  Serogroup C | 97.7 [94.3 to 99.4] | 98.9 [93.8 to 100.0] | 100.0 [97.6 to 100] | 98.7 [93.1 to 100.0] | 90.8 [85.9 to 94.5] | 91.7 [84.2 to 96.3]
  Serogroup Y | 93.2 [88.5 to 96.4] | 88.5 [79.9 to 94.3] | 92.3 [86.9 to 95.9] | 87.3 [78.0 to 93.8] | 92.9 [88.3 to 96.0] | 92.7 [85.6 to 97.0]
  Serogroup W | 86.4 [80.5 to 91.1] | 83.9 [74.5 to 90.9] | 82.6 [75.7 to 88.2] | 82.3 [72.1 to 90.0] | 82.1 [76.1 to 87.2] | 90.6 [82.9 to 95.6]

5. Secondary Outcome: Geometric Mean Titers of MMR-Varicella Antibodies Following Injection With MMR-Varicella Vaccine Administered Alone or Concomitantly With the MenACYW Conjugate Vaccine: Groups 1, 3, 10, and 12
Description: Antibodies titers of Measles and Rubella were measured by enzyme immunoassay (EIA). Antibodies titers for mumps and varicella were measured by enzyme-linked immunosorbent assay (ELISA). Data for this outcome measure was planned to be reported for the combined population of Groups 1 and 10, Groups 3 and 12.
Time Frame: Day 0 and Day 30 post-vaccination
Population: Analysis was performed on PPAS. Here, 'Number analyzed' = participants with available data for each specified category. Data for this outcome measure were not planned to be collected and analyzed for Groups 2, 4, 5, 6, 7, 8, 9, and 11.
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Groups:
- Groups 3 and 12: MMR + Varicella Vaccine: Healthy, meningococcal-vaccine naïve toddlers (aged 12 to 23 months) from South Korea and Thailand received single dose of MMR vaccine and varicella vaccine on Day 0.
Arm/Group | Groups 1 and10:MenACYW Conjugate Vaccine+MMR+Varicella Vaccine | Groups 3 and 12: MMR + Varicella Vaccine
Number analyzed (Participants) | 177 | 92
titers (1/dilution)
  Measles: Day 0: number analyzed (Participants) | 176 | 92
  Measles: Day 0 | 40.0 [37.2 to 43.1] | 45.0 [40.1 to 50.4]
  Measles: Day 30 | 2156 [1893 to 2455] | 2840 [2389 to 3378]
  Mumps: Day 0: number analyzed (Participants) | 176 | 92
  Mumps: Day 0 | 5.51 [5.20 to 5.84] | 5.43 [5.05 to 5.83]
  Mumps: Day 30 | 85.9 [74.7 to 98.7] | 97.6 [83.1 to 115]
  Rubella: Day 0: number analyzed (Participants) | 176 | 92
  Rubella: Day 0 | 5.94 [5.32 to 6.63] | 7.12 [6.07 to 8.34]
  Rubella: Day 30 | 87.6 [79.4 to 96.7] | 104 [91.2 to 118]
  Varicella: Day 0: number analyzed (Participants) | 176 | 92
  Varicella: Day 0 | 0.556 [0.484 to 0.638] | 0.665 [0.508 to 0.869]
  Varicella: Day 30 | 13.4 [11.6 to 15.4] | 17.4 [15.2 to 19.9]

6. Secondary Outcome: Percentage of Participants With Immune Response Following Injection With MMR-Varicella Vaccine Administered Alone or Concomitantly With the MenACYW Conjugate Vaccine: Groups 1, 3, 10, and 12
Description: Immune response for MMR-Varicella vaccine was defined as: anti-measles Antibody (Ab) concentrations >=255 milli-international unit per milliliter (mIU/mL), anti-mumps Ab concentrations: >=10 Ab units/mL, anti-rubella Ab concentrations >=10 international unit per milliliter (IU/mL),anti-varicella Ab concentrations >=5 glycoprotein enzyme-linked immunosorbent assay (gpELISA) Ab units/mL. Data for this outcome measure was planned to be reported for the combined population of Groups 1 and 10, Groups 3 and 12.
Time Frame: Day 0 and Day 30 post-vaccination
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Groups 1 and10:MenACYW Conjugate Vaccine+MMR+Varicella Vaccine | Groups 3 and 12: MMR + Varicella Vaccine
Number analyzed (Participants) | 177 | 92
percentage of participants
  Measles: Day 0: number analyzed (Participants) | 176 | 92
  Measles: Day 0 | 0.6 [0.0 to 3.1] | 0.0 [0.0 to 3.9]
  Measles: Day 30 | 96.6 [92.8 to 98.7] | 97.8 [92.4 to 99.7]
  Mumps: Day 0: number analyzed (Participants) | 176 | 92
  Mumps: Day 0 | 7.4 [4.0 to 12.3] | 6.5 [2.4 to 13.7]
  Mumps: Day 30 | 97.7 [94.3 to 99.4] | 100.0 [96.1 to 100.0]
  Rubella: Day 0: number analyzed (Participants) | 176 | 92
  Rubella: Day 0 | 27.3 [20.8 to 34.5] | 31.5 [22.2 to 42.0]
  Rubella: Day 30 | 100.0 [97.9 to 100] | 100.0 [96.1 to 100]
  Varicella: Day 0: number analyzed (Participants) | 176 | 92
  Varicella: Day 0 | 4.0 [1.6 to 8.0] | 7.6 [3.1 to 15.1]
  Varicella: Day 30 | 93.2 [88.5 to 96.4] | 98.9 [94.1 to 100.0]

7. Secondary Outcome: Geometric Mean Titers of Pertussis Toxoid (PT) and Filamentous Hemagglutinin (FHA) Antibodies Following Injection With DTaP-IPV-HB-Hib Vaccine Administrated Alone or Concomitantly With the MenACYW Conjugate Vaccine: Groups 4 and 6
Description: Antibodies titers of PT and FHA were measured by electrochemiluminescent (ECL) assay.
Time Frame: Day 0 and Day 30 post-vaccination
Population: Analysis was performed on PPAS. Data for this outcome measure were not planned to be collected and analyzed for Groups 1, 2, 3, 5, 7, 8, 9, 10, 11, and 12.
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | Mexico (Group 4): MenACYW Conjugate + DTaP-IPV-HB-Hib Vaccine | Mexico (Group 6): DTaP-IPV-HB-Hib Vaccine
Number analyzed (Participants) | 155 | 68
titers (1/dilution)
  PT: Day 0 | 17.9 [15.1 to 21.3] | 20.4 [15.3 to 27.0]
  PT: Day 30 | 144 [130 to 159] | 169 [144 to 198]
  FHA: Day 0 | 45.5 [37.0 to 55.9] | 57.4 [41.4 to 79.5]
  FHA: Day 30 | 299 [265 to 337] | 391 [319 to 480]

8. Secondary Outcome: Geometric Mean Titers of DTaP-IPV-HB-Hib Antibodies Following Injection With DTaP-IPV-HB-Hib Administered Alone or Concomitantly With the MenACYW Conjugate Vaccine: Groups 4 and 6
Description: Antibodies titers of Diphtheria, Tetanus and Pertussis were measured by ECL assay. Antibodies titers of poliovirus types 1, 2, and 3 were measured by neutralization assay. Antibodies titers of Hepatitis B were measured by an immunodiagnostic system using chemiluminescence detection. Antibodies titers of Polyribosyl-ribitol phosphate (PRP) were measured by Farr-type radioimmunoassay (RIA).
Time Frame: Day 0 (for tetanus only) and Day 30 post-vaccination
Population: Analysis was performed on PPAS. Here, 'Number analyzed' = participants with available data for each specified category. Data for this outcome measure were not planned to be collected and analyzed for Groups 1, 2, 3, 5, 7, 8, 9, 10, 11, and 12.
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | Mexico (Group 4): MenACYW Conjugate + DTaP-IPV-HB-Hib Vaccine | Mexico (Group 6): DTaP-IPV-HB-Hib Vaccine
Number analyzed (Participants) | 155 | 68
titers (1/dilution)
  Diphtheria: Day 30 | 5.52 [4.94 to 6.17] | 6.34 [5.51 to 7.30]
  Tetanus: Day 0: number analyzed (Participants) | 155 | 67
  Tetanus: Day 0 | 0.238 [0.196 to 0.289] | 0.234 [0.177 to 0.309]
  Tetanus: Day 30 | 7.06 [6.01 to 8.29] | 7.11 [5.79 to 8.74]
  Polio 1: Day 30 | 4560 [3870 to 5373] | 4034 [3052 to 5332]
  Polio 2: Day 30 | 7244 [6208 to 8453] | 5618 [4578 to 6895]
  Polio 3: Day 30 | 5977 [4958 to 7205] | 5100 [3840 to 6772]
  Hepatitis B: Day 30 | 5171 [4104 to 6515] | 7308 [5135 to 10401]
  PRP: Day 30 | 46.6 [39.6 to 54.9] | 56.2 [41.5 to 76.1]

9. Secondary Outcome: Percentage of Participants With Immune Response Following Injection With DTaP-IPV-HB-Hib Vaccine Administered Alone or Concomitantly With the MenACYW Conjugate Vaccine: Groups 4 and 6
Description: Immune response for DTaP-IPV-HB-Hib vaccine was defined as: anti-tetanus Ab concentrations: >= 0.01 and 0.1 IU/mL at Day 0 and >= 0.1 and 1.0 IU/mL at Day 30, anti-diphtheria Ab concentrations: >= 0.1 and 1.0 IU/mL, anti-PRP Ab concentrations >= 0.15 and 1.0 microgram per milliliter (mcg/mL), anti-poliovirus types 1, 2, and 3 Ab titers >= 1:8, anti-hepatitis B surface antigen Ab concentrations >= 10 mIU/mL, >= 100 mIU/mL.
Time Frame: Day 0 (tetanus only) and Day 30 post-vaccination
Population: Analysis was performed on PPAS. Here, 'Number analyzed' = participants with available data for each specified category. Data for this outcome measure were not planned to be collected and analyzed for Groups 1, 2, 3, 5, 7, 8, 9, 10, 11 and 12.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Mexico (Group 4): MenACYW Conjugate + DTaP-IPV-HB-Hib Vaccine: Healthy, meningococcal-vaccine naïve toddlers (aged 12 to 23 months) received single dose of MenACYW Conjugate and DTaP-IPV-HB-Hib vaccine on Day 0.
Arm/Group | Mexico (Group 4): MenACYW Conjugate + DTaP-IPV-HB-Hib Vaccine | Mexico (Group 6): DTaP-IPV-HB-Hib Vaccine
Number analyzed (Participants) | 155 | 68
percentage of participants
  Diphtheria: Day 30 (>=0.1 IU/mL) | 100.0 [97.6 to 100] | 100.0 [94.7 to 100]
  Diphtheria: Day 30 (>=1 IU/mL) | 98.7 [95.4 to 99.8] | 100.0 [94.7 to 100]
  Tetanus: Day 0 (>=0.01 IU/mL): number analyzed (Participants) | 155 | 67
  Tetanus: Day 0 (>=0.01 IU/mL) | 100.0 [97.6 to 100] | 100.0 [94.6 to 100]
  Tetanus: Day 0 (>=0.1 IU/mL): number analyzed (Participants) | 155 | 67
  Tetanus: Day 0 (>=0.1 IU/mL) | 81.3 [74.2 to 87.1] | 77.6 [65.8 to 86.9]
  Tetanus: Day 30 (>=0.1 IU/mL) | 100.0 [97.6 to 100] | 100.0 [94.7 to 100]
  Tetanus: Day 30 (>=1 IU/mL) | 98.1 [94.4 to 99.6] | 98.5 [92.1 to 100.0]
  Polio 1: Day 30 (>=8 [1/dilution]) | 100.0 [97.6 to 100] | 100.0 [94.7 to 100]
  Polio 2: Day 30 (>=8 [1/dilution]) | 100.0 [97.6 to 100] | 100.0 [94.7 to 100]
  Polio 3: Day 30 (>=8 [1/dilution]) | 100.0 [97.6 to 100] | 100.0 [94.7 to 100]
  Hepatitis B: Day 30 (>=10 mIU/mL) | 100.0 [97.6 to 100] | 100.0 [94.7 to 100]
  Hepatitis B: Day 30 (>=100 mIU/mL) | 98.7 [95.4 to 99.8] | 100.0 [94.7 to 100]
  PRP: Day 30 (>=0.15 mcg/mL) | 100.0 [97.6 to 100] | 100.0 [94.7 to 100]
  PRP: Day 30 (>=1.0 mcg/mL) | 100.0 [97.6 to 100] | 100.0 [94.7 to 100]

10. Secondary Outcome: Percentage of Participants With Vaccine Response of PT and FHA Antibodies Following Injection With DTaP-IPV-HB-Hib Vaccine Administered Alone or Concomitantly With the MenACYW Conjugate Vaccine: Groups 4 and 6
Description: Pertussis and FHA vaccine response was defined as: if the pre-vaccination concentration is < 4 * lower limit of quantification (LLOQ is equal to 2), then the post-vaccination concentration is >=4 * pre-vaccination concentration and if the pre-vaccination concentration is >= 4 * LLOQ, then the post-vaccination concentration is >= 2 * pre-vaccination concentration.
Time Frame: Day 0 and Day 30 post-vaccination
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mexico (Group 4): MenACYW Conjugate + DTaP-IPV-HB-Hib Vaccine | Mexico (Group 6): DTaP-IPV-HB-Hib Vaccine
Number analyzed (Participants) | 155 | 68
percentage of participants
  PT: Day 30/Day 0 | 91.0 [85.3 to 95.0] | 92.6 [83.7 to 97.6]
  FHA: Day 30/Day 0 | 89.0 [83.0 to 93.5] | 88.2 [78.1 to 94.8]

11. Secondary Outcome: Geometric Mean Titers of PCV13 Serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F Antibodies Following Injection With PCV13 Vaccine Administrated Alone or Concomitantly With the MenACYW Conjugate Vaccine: Groups 7 and 9
Description: Antibodies of pneumococcal serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F were measured by ECL assay.
Time Frame: Day 0 and Day 30 post-vaccination
Population: Analysis was performed on PPAS. Here, 'Number analyzed' = participants with available data for each specified category. Data for this outcome measure were not planned to be collected and analyzed for Groups 1, 2, 3, 4, 5, 6, 8, 10, 11, and 12.
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Groups:
- Russian Federation (Group 7):MenACYW Conjugate + PCV13 Vaccine: Healthy, meningococcal-vaccine naïve toddlers (aged 15 to 23 months) received single dose of MenACYW Conjugate vaccine and PCV13 vaccine on Day 0.
Arm/Group | Russian Federation (Group 7):MenACYW Conjugate + PCV13 Vaccine | Russian Federation (Group 9): PCV13 Vaccine
Number analyzed (Participants) | 196 | 92
titers (1/dilution)
  Serotype 1: Day 0: number analyzed (Participants) | 193 | 92
  Serotype 1: Day 0 | 0.867 [0.741 to 1.01] | 0.918 [0.713 to 1.18]
  Serotype 1: Day 30: number analyzed (Participants) | 191 | 92
  Serotype 1: Day 30 | 2.33 [1.98 to 2.75] | 2.14 [1.63 to 2.81]
  Serotype 3: Day 0: number analyzed (Participants) | 193 | 92
  Serotype 3: Day 0 | 0.409 [0.341 to 0.491] | 0.414 [0.322 to 0.533]
  Serotype 3: Day 30: number analyzed (Participants) | 191 | 92
  Serotype 3: Day 30 | 0.802 [0.664 to 0.967] | 0.773 [0.608 to 0.983]
  Serotype 4: Day 0: number analyzed (Participants) | 193 | 92
  Serotype 4: Day 0 | 0.604 [0.511 to 0.715] | 0.653 [0.507 to 0.840]
  Serotype 4: Day 30: number analyzed (Participants) | 191 | 92
  Serotype 4: Day 30 | 1.97 [1.68 to 2.31] | 1.49 [1.15 to 1.93]
  Serotype 5: Day 0: number analyzed (Participants) | 193 | 92
  Serotype 5: Day 0 | 0.828 [0.719 to 0.953] | 0.782 [0.610 to 1.00]
  Serotype 5: Day 30: number analyzed (Participants) | 191 | 92
  Serotype 5: Day 30 | 1.99 [1.70 to 2.31] | 1.73 [1.33 to 2.24]
  Serotype 6A: Day 0: number analyzed (Participants) | 193 | 92
  Serotype 6A: Day 0 | 1.61 [1.33 to 1.95] | 1.48 [1.09 to 2.00]
  Serotype 6A: Day 30: number analyzed (Participants) | 191 | 92
  Serotype 6A: Day 30 | 5.96 [4.99 to 7.13] | 6.13 [4.47 to 8.41]
  Serotype 6B: Day 0: number analyzed (Participants) | 193 | 92
  Serotype 6B: Day 0 | 0.895 [0.715 to 1.12] | 0.691 [0.514 to 0.929]
  Serotype 6B: Day 30: number analyzed (Participants) | 191 | 92
  Serotype 6B: Day 30 | 3.66 [2.99 to 4.50] | 2.57 [1.83 to 3.61]
  Serotype 7F: Day 0: number analyzed (Participants) | 193 | 92
  Serotype 7F: Day 0 | 1.32 [1.12 to 1.55] | 1.39 [1.08 to 1.77]
  Serotype 7F: Day 30: number analyzed (Participants) | 191 | 92
  Serotype 7F: Day 30 | 3.05 [2.59 to 3.58] | 2.67 [2.05 to 3.47]
  Serotype 9V: Day 0: number analyzed (Participants) | 193 | 92
  Serotype 9V: Day 0 | 0.841 [0.710 to 0.997] | 0.863 [0.660 to 1.13]
  Serotype 9V: Day 30: number analyzed (Participants) | 191 | 92
  Serotype 9V: Day 30 | 2.34 [1.95 to 2.81] | 2.52 [1.92 to 3.30]
  Serotype 14: Day 0: number analyzed (Participants) | 192 | 92
  Serotype 14: Day 0 | 3.25 [2.74 to 3.86] | 3.00 [2.30 to 3.91]
  Serotype 14: Day 30: number analyzed (Participants) | 191 | 92
  Serotype 14: Day 30 | 7.62 [6.56 to 8.83] | 6.30 [5.00 to 7.93]
  Serotype 18C: Day 0: number analyzed (Participants) | 193 | 92
  Serotype 18C: Day 0 | 0.737 [0.620 to 0.876] | 0.995 [0.766 to 1.29]
  Serotype 18C: Day 30: number analyzed (Participants) | 191 | 92
  Serotype 18C: Day 30 | 2.19 [1.87 to 2.58] | 2.21 [1.73 to 2.83]
  Serotype 19A: Day 0: number analyzed (Participants) | 193 | 92
  Serotype 19A: Day 0 | 1.65 [1.36 to 2.01] | 1.96 [1.46 to 2.64]
  Serotype 19A: Day 30: number analyzed (Participants) | 191 | 92
  Serotype 19A: Day 30 | 5.75 [4.85 to 6.80] | 5.91 [4.54 to 7.69]
  Serotype 19F: Day 0: number analyzed (Participants) | 193 | 92
  Serotype 19F: Day 0 | 1.78 [1.43 to 2.21] | 1.74 [1.28 to 2.35]
  Serotype 19F: Day 30: number analyzed (Participants) | 191 | 92
  Serotype 19F: Day 30 | 5.58 [4.57 to 6.81] | 5.53 [3.98 to 7.69]
  Serotype 23F: Day 0: number analyzed (Participants) | 192 | 92
  Serotype 23F: Day 0 | 0.631 [0.519 to 0.768] | 0.733 [0.537 to 1.00]
  Serotype 23F: Day 30: number analyzed (Participants) | 191 | 92
  Serotype 23F: Day 30 | 2.42 [2.04 to 2.86] | 2.58 [1.98 to 3.37]

12. Secondary Outcome: Percentage of Participants With Immune Response Following Injection With PCV13 Vaccine Administered Alone or Concomitantly With the MenACYW Conjugate Vaccine: Groups 7 and 9
Description: Immune response for PCV13 for serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F was defined as: antibodies concentrations >=0.35 mcg/mL or >=1.0 mcg/mL.
Time Frame: Day 0 and Day 30 post-vaccination
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Russian Federation (Group 7):MenACYW Conjugate + PCV13 Vaccine | Russian Federation (Group 9): PCV13 Vaccine
Number analyzed (Participants) | 196 | 92
percentage of participants
  Serotype 1: Day 0 (>=0.35 mcg/mL): number analyzed (Participants) | 193 | 92
  Serotype 1: Day 0 (>=0.35 mcg/mL) | 80.8 [74.6 to 86.1] | 79.3 [69.6 to 87.1]
  Serotype 1: Day 0 (>=1.0 mcg/mL): number analyzed (Participants) | 193 | 92
  Serotype 1: Day 0 (>=1.0 mcg/mL) | 43.0 [35.9 to 50.3] | 45.7 [35.2 to 56.4]
  Serotype 1: Day 30 (>=0.35 mcg/mL): number analyzed (Participants) | 191 | 92
  Serotype 1: Day 30 (>=0.35 mcg/mL) | 97.4 [94.0 to 99.1] | 94.6 [87.8 to 98.2]
  Serotype 1: Day 30 (>=1.0 mcg/mL): number analyzed (Participants) | 191 | 92
  Serotype 1: Day 30 (>=1.0 mcg/mL) | 76.4 [69.8 to 82.3] | 70.7 [60.2 to 79.7]
  Serotype 3: Day 0 (>=0.35 mcg/mL): number analyzed (Participants) | 193 | 92
  Serotype 3: Day 0 (>=0.35 mcg/mL) | 49.2 [42.0 to 56.5] | 53.3 [42.6 to 63.7]
  Serotype 3: Day 0 (>=1.0 mcg/mL): number analyzed (Participants) | 193 | 92
  Serotype 3: Day 0 (>=1.0 mcg/mL) | 22.3 [16.6 to 28.8] | 18.5 [11.1 to 27.9]
  Serotype 3: Day 30 (>=0.35 mcg/mL): number analyzed (Participants) | 191 | 92
  Serotype 3: Day 30 (>=0.35 mcg/mL) | 72.3 [65.3 to 78.5] | 76.1 [66.1 to 84.4]
  Serotype 3: Day 30 (>=1.0 mcg/mL): number analyzed (Participants) | 191 | 92
  Serotype 3: Day 30 (>=1.0 mcg/mL) | 48.2 [40.9 to 55.5] | 38.0 [28.1 to 48.8]
  Serotype 4: Day 0 (>=0.35 mcg/mL): number analyzed (Participants) | 193 | 92
  Serotype 4: Day 0 (>=0.35 mcg/mL) | 66.8 [59.7 to 73.4] | 68.5 [58.0 to 77.8]
  Serotype 4: Day 0 (>=1.0 mcg/mL): number analyzed (Participants) | 193 | 92
  Serotype 4: Day 0 (>=1.0 mcg/mL) | 33.7 [27.1 to 40.8] | 38.0 [28.1 to 48.8]
  Serotype 4: Day 30 (>=0.35 mcg/mL): number analyzed (Participants) | 191 | 92
  Serotype 4: Day 30 (>=0.35 mcg/mL) | 92.7 [88.0 to 95.9] | 90.2 [82.2 to 95.4]
  Serotype 4: Day 30 (>=1.0 mcg/mL): number analyzed (Participants) | 191 | 92
  Serotype 4: Day 30 (>=1.0 mcg/mL) | 80.1 [73.7 to 85.5] | 62.0 [51.2 to 71.9]
  Serotype 5: Day 0 (>=0.35 mcg/mL): number analyzed (Participants) | 193 | 92
  Serotype 5: Day 0 (>=0.35 mcg/mL) | 81.3 [75.1 to 86.6] | 76.1 [66.1 to 84.4]
  Serotype 5: Day 0 (>=1.0 mcg/mL): number analyzed (Participants) | 193 | 92
  Serotype 5: Day 0 (>=1.0 mcg/mL) | 41.5 [34.4 to 48.7] | 50.0 [39.4 to 60.6]
  Serotype 5: Day 30 (>=0.35 mcg/mL): number analyzed (Participants) | 191 | 92
  Serotype 5: Day 30 (>=0.35 mcg/mL) | 94.8 [90.6 to 97.5] | 90.2 [82.2 to 95.4]
  Serotype 5: Day 30 (>=1.0 mcg/mL): number analyzed (Participants) | 191 | 92
  Serotype 5: Day 30 (>=1.0 mcg/mL) | 71.2 [64.2 to 77.5] | 69.6 [59.1 to 78.7]
  Serotype 6A: Day 0 (>=0.35 mcg/mL): number analyzed (Participants) | 193 | 92
  Serotype 6A: Day 0 (>=0.35 mcg/mL) | 90.2 [85.1 to 94.0] | 82.6 [73.3 to 89.7]
  Serotype 6A: Day 0 (>=1.0 mcg/mL): number analyzed (Participants) | 193 | 92
  Serotype 6A: Day 0 (>=1.0 mcg/mL) | 63.7 [56.5 to 70.5] | 65.2 [54.6 to 74.9]
  Serotype 6A: Day 30 (>=0.35 mcg/mL): number analyzed (Participants) | 191 | 92
  Serotype 6A: Day 30 (>=0.35 mcg/mL) | 97.4 [94.0 to 99.1] | 96.7 [90.8 to 99.3]
  Serotype 6A: Day 30 (>=1.0 mcg/mL): number analyzed (Participants) | 191 | 92
  Serotype 6A: Day 30 (>=1.0 mcg/mL) | 96.3 [92.6 to 98.5] | 90.2 [82.2 to 95.4]
  Serotype 6B: Day 0 (>=0.35 mcg/mL): number analyzed (Participants) | 193 | 92
  Serotype 6B: Day 0 (>=0.35 mcg/mL) | 72.0 [65.1 to 78.2] | 68.5 [58.0 to 77.8]
  Serotype 6B: Day 0 (>=1.0 mcg/mL): number analyzed (Participants) | 193 | 92
  Serotype 6B: Day 0 (>=1.0 mcg/mL) | 44.6 [37.4 to 51.9] | 41.3 [31.1 to 52.1]
  Serotype 6B: Day 30 (>=0.35 mcg/mL): number analyzed (Participants) | 191 | 92
  Serotype 6B: Day 30 (>=0.35 mcg/mL) | 94.8 [90.6 to 97.5] | 92.4 [84.9 to 96.9]
  Serotype 6B: Day 30 (>=1.0 mcg/mL): number analyzed (Participants) | 191 | 92
  Serotype 6B: Day 30 (>=1.0 mcg/mL) | 86.4 [80.7 to 90.9] | 75.0 [64.9 to 83.4]
  Serotype 7F: Day 0 (>=0.35 mcg/mL): number analyzed (Participants) | 193 | 92
  Serotype 7F: Day 0 (>=0.35 mcg/mL) | 87.0 [81.5 to 91.4] | 88.0 [79.6 to 93.9]
  Serotype 7F: Day 0 (>=1.0 mcg/mL): number analyzed (Participants) | 193 | 92
  Serotype 7F: Day 0 (>=1.0 mcg/mL) | 62.7 [55.5 to 69.5] | 65.2 [54.6 to 74.9]
  Serotype 7F: Day 30 (>=0.35 mcg/mL): number analyzed (Participants) | 191 | 92
  Serotype 7F: Day 30 (>=0.35 mcg/mL) | 98.4 [95.5 to 99.7] | 94.6 [87.8 to 98.2]
  Serotype 7F: Day 30 (>=1.0 mcg/mL): number analyzed (Participants) | 191 | 92
  Serotype 7F: Day 30 (>=1.0 mcg/mL) | 80.1 [73.7 to 85.5] | 83.7 [74.5 to 90.6]
  Serotype 9V: Day 0 (>=0.35 mcg/mL): number analyzed (Participants) | 193 | 92
  Serotype 9V: Day 0 (>=0.35 mcg/mL) | 77.2 [70.6 to 82.9] | 79.3 [69.6 to 87.1]
  Serotype 9V: Day 0 (>=1.0 mcg/mL): number analyzed (Participants) | 193 | 92
  Serotype 9V: Day 0 (>=1.0 mcg/mL) | 42.0 [34.9 to 49.3] | 43.5 [33.2 to 54.2]
  Serotype 9V: Day 30 (>=0.35 mcg/mL): number analyzed (Participants) | 191 | 92
  Serotype 9V: Day 30 (>=0.35 mcg/mL) | 95.3 [91.2 to 97.8] | 92.4 [84.9 to 96.9]
  Serotype 9V: Day 30 (>=1.0 microg/mL): number analyzed (Participants) | 191 | 92
  Serotype 9V: Day 30 (>=1.0 microg/mL) | 74.3 [67.5 to 80.4] | 75.0 [64.9 to 83.4]
  Serotype 14: Day 0 (>=0.35 mcg/mL): number analyzed (Participants) | 192 | 92
  Serotype 14: Day 0 (>=0.35 mcg/mL) | 95.8 [92.0 to 98.2] | 92.4 [84.9 to 96.9]
  Serotype 14: Day 0 (>=1.0 mcg/mL): number analyzed (Participants) | 192 | 92
  Serotype 14: Day 0 (>=1.0 mcg/mL) | 83.3 [77.3 to 88.3] | 87.0 [78.3 to 93.1]
  Serotype 14: Day 30 (>=0.35 mcg/mL): number analyzed (Participants) | 191 | 92
  Serotype 14: Day 30 (>=0.35 mcg/mL) | 99.0 [96.3 to 99.9] | 98.9 [94.1 to 100.0]
  Serotype 14: Day 30 (>=1.0 mcg/mL): number analyzed (Participants) | 191 | 92
  Serotype 14: Day 30 (>=1.0 mcg/mL) | 97.4 [94.0 to 99.1] | 94.6 [87.8 to 98.2]
  Serotype 18C: Day 0 (>=0.35 mcg/mL): number analyzed (Participants) | 193 | 92
  Serotype 18C: Day 0 (>=0.35 mcg/mL) | 71.5 [64.6 to 77.8] | 84.8 [75.8 to 91.4]
  Serotype 18C: Day 0 (>=1.0 mcg/mL): number analyzed (Participants) | 193 | 92
  Serotype 18C: Day 0 (>=1.0 mcg/mL) | 40.9 [33.9 to 48.2] | 48.9 [38.3 to 59.6]
  Serotype 18C: Day 30 (>=0.35 mcg/mL): number analyzed (Participants) | 191 | 92
  Serotype 18C: Day 30 (>=0.35 mcg/mL) | 95.3 [91.2 to 97.8] | 92.4 [84.9 to 96.9]
  Serotype 18C: Day 30 (>=1.0 mcg/mL): number analyzed (Participants) | 191 | 92
  Serotype 18C: Day 30 (>=1.0 mcg/mL) | 79.1 [72.6 to 84.6] | 79.3 [69.6 to 87.1]
  Serotype 19A: Day 0 (>=0.35 mcg/mL): number analyzed (Participants) | 193 | 92
  Serotype 19A: Day 0 (>=0.35 mcg/mL) | 87.0 [81.5 to 91.4] | 87.0 [78.3 to 93.1]
  Serotype 19A: Day 0 (>=1.0 mcg/mL): number analyzed (Participants) | 193 | 92
  Serotype 19A: Day 0 (>=1.0 mcg/mL) | 62.7 [55.5 to 69.5] | 69.6 [59.1 to 78.7]
  Serotype 19A: Day 30 (>=0.35 mcg/mL): number analyzed (Participants) | 191 | 92
  Serotype 19A: Day 30 (>=0.35 mcg/mL) | 96.3 [92.6 to 98.5] | 98.9 [94.1 to 100.0]
  Serotype 19A: Day 30 (>=1.0 mcg/mL): number analyzed (Participants) | 191 | 92
  Serotype 19A: Day 30 (>=1.0 mcg/mL) | 92.7 [88.0 to 95.9] | 90.2 [82.2 to 95.4]
  Serotype 19F: Day 0 (>=0.35 mcg/mL): number analyzed (Participants) | 193 | 92
  Serotype 19F: Day 0 (>=0.35 mcg/mL) | 87.0 [81.5 to 91.4] | 89.1 [80.9 to 94.7]
  Serotype 19F: Day 0 (>=1.0 mcg/mL): number analyzed (Participants) | 193 | 92
  Serotype 19F: Day 0 (>=1.0 mcg/mL) | 64.2 [57.0 to 71.0] | 65.2 [54.6 to 74.9]
  Serotype 19F: Day 30 (>=0.35 mcg/mL): number analyzed (Participants) | 191 | 92
  Serotype 19F: Day 30 (>=0.35 mcg/mL) | 96.9 [93.3 to 98.8] | 97.8 [92.4 to 99.7]
  Serotype 19F: Day 30 (>=1.0 mcg/mL): number analyzed (Participants) | 191 | 92
  Serotype 19F: Day 30 (>=1.0 mcg/mL) | 88.0 [82.5 to 92.2] | 85.9 [77.0 to 92.3]
  Serotype 23F: Day 0 (>=0.35 mcg/mL): number analyzed (Participants) | 192 | 92
  Serotype 23F: Day 0 (>=0.35 mcg/mL) | 68.2 [61.1 to 74.7] | 64.1 [53.5 to 73.9]
  Serotype 23F: Day 0 (>=1.0 mcg/mL): number analyzed (Participants) | 192 | 92
  Serotype 23F: Day 0 (>=1.0 mcg/mL) | 34.9 [28.2 to 42.1] | 44.6 [34.2 to 55.3]
  Serotype 23F: Day 30 (>=0.35 mcg/mL): number analyzed (Participants) | 191 | 92
  Serotype 23F: Day 30 (>=0.35 mcg/mL) | 96.3 [92.6 to 98.5] | 93.5 [86.3 to 97.6]
  Serotype 23F: Day 30 (>=1.0 mcg/mL): number analyzed (Participants) | 191 | 92
  Serotype 23F: Day 30 (>=1.0 mcg/mL) | 72.3 [65.3 to 78.5] | 78.3 [68.4 to 86.2]

13. Secondary Outcome: Number of Participants Reporting at Least One Solicited Injection Site Reactions (Tenderness, Erythema, and Swelling): Groups 1, 2, 3, 10, 11, and 12
Description: Solicited Reaction (SR) was defined as an adverse event (AE) that was prelisted (i.e., solicited) in the electronic case report form (eCRF) and considered to be related to vaccination (adverse drug reaction). Solicited injection site reactions: tenderness, erythema, and swelling. Tenderness: Grade 3: cries when injected limb moved or the movement of the injected limb reduced, Erythema and swelling: Grade 3: >= 50 millimeter (mm). Participants with any of the Grade and Grade 3 solicited injection-site reactions were reported.
Time Frame: Within 7 days post vaccination
Population: Analysis was performed on Safety analysis set (SafAS) which included participants who received at least 1 dose of study vaccine(s) & had any safety data available. Here '0' in the number analyzed field signifies that the vaccines mentioned in the respective categories were not administered to the specified group.
Measure: Count of Participants; unit: Participants
Groups:
- South Korea(Group1):MenACYW Conjugate +MMR +Varicella Vaccine: Healthy, meningococcal-vaccine naïve toddlers (aged 12 to 23 months) received single dose MenACYW Conjugate vaccine, MMR vaccine, and varicella vaccine on Day 0.
- Thailand (Group 10):MenACYW Conjugate + MMR +Varicella Vaccine: Healthy, meningococcal-vaccine naïve toddlers (aged 12 to 23 months) received single dose of MenACYW Conjugate vaccine, MMR vaccine, and varicella vaccine on Day 0.
- Thailand (Group 12): MMR +Varicella Vaccine: Healthy, meningococcal-vaccine naïve toddlers (aged 12 to 23 months) received single dose of MMR vaccine and varicella vaccine on Day 0.
Arm/Group | South Korea(Group1):MenACYW Conjugate +MMR +Varicella Vaccine | South Korea (Group 2): MenACYW Conjugate Vaccine | South Korea (Group 3): MMR + Varicella Vaccine | Thailand (Group 10):MenACYW Conjugate + MMR +Varicella Vaccine | Thailand (Group 11): MenACYW Conjugate Vaccine | Thailand (Group 12): MMR +Varicella Vaccine
Number analyzed (Participants) | 103 | 52 | 53 | 86 | 42 | 42
Participants
  MenACYW: Tenderness: Any Grade: number analyzed (Participants) | 103 | 52 | 0 | 86 | 42 | 0
  MenACYW: Tenderness: Any Grade | 28 | 15 |  | 29 | 17 |
  MenACYW: Tenderness: Grade 3: number analyzed (Participants) | 103 | 52 | 0 | 86 | 42 | 0
  MenACYW: Tenderness: Grade 3 | 1 | 0 |  | 0 | 1 |
  MenACYW: Erythema: Any Grade: number analyzed (Participants) | 103 | 52 | 0 | 86 | 42 | 0
  MenACYW: Erythema: Any Grade | 27 | 20 |  | 29 | 13 |
  MenACYW: Erythema: Grade 3: number analyzed (Participants) | 103 | 52 | 0 | 86 | 42 | 0
  MenACYW: Erythema: Grade 3 | 0 | 2 |  | 0 | 0 |
  MenACYW: Swelling: Any Grade: number analyzed (Participants) | 103 | 52 | 0 | 86 | 42 | 0
  MenACYW: Swelling: Any Grade | 18 | 14 |  | 15 | 7 |
  MenACYW: Swelling: Grade 3: number analyzed (Participants) | 103 | 52 | 0 | 86 | 42 | 0
  MenACYW: Swelling: Grade 3 | 0 | 0 |  | 0 | 0 |
  MMR: Tenderness: Any Grade: number analyzed (Participants) | 103 | 0 | 53 | 86 | 0 | 42
  MMR: Tenderness: Any Grade | 21 |  | 10 | 17 |  | 18
  MMR: Tenderness: Grade 3: number analyzed (Participants) | 103 | 0 | 53 | 86 | 0 | 42
  MMR: Tenderness: Grade 3 | 1 |  | 0 | 0 |  | 0
  MMR: Erythema: Any Grade: number analyzed (Participants) | 103 | 0 | 53 | 86 | 0 | 42
  MMR: Erythema: Any Grade | 13 |  | 6 | 24 |  | 10
  MMR: Erythema: Grade 3: number analyzed (Participants) | 103 | 0 | 53 | 86 | 0 | 42
  MMR: Erythema: Grade 3 | 0 |  | 0 | 0 |  | 0
  MMR: Swelling: Any Grade: number analyzed (Participants) | 103 | 0 | 53 | 86 | 0 | 42
  MMR: Swelling: Any Grade | 7 |  | 1 | 11 |  | 4
  MMR: Swelling: Grade 3: number analyzed (Participants) | 103 | 0 | 53 | 86 | 0 | 42
  MMR: Swelling: Grade 3 | 0 |  | 0 | 0 |  | 0
  Varicella: Tenderness: Any Grade: number analyzed (Participants) | 103 | 0 | 53 | 86 | 0 | 42
  Varicella: Tenderness: Any Grade | 23 |  | 11 | 17 |  | 14
  Varicella: Tenderness: Grade 3: number analyzed (Participants) | 103 | 0 | 53 | 86 | 0 | 42
  Varicella: Tenderness: Grade 3 | 0 |  | 0 | 0 |  | 1
  Varicella: Erythema: Any Grade: number analyzed (Participants) | 103 | 0 | 53 | 86 | 0 | 42
  Varicella: Erythema: Any Grade | 19 |  | 4 | 18 |  | 13
  Varicella: Erythema: Grade 3: number analyzed (Participants) | 103 | 0 | 53 | 86 | 0 | 42
  Varicella: Erythema: Grade 3 | 1 |  | 0 | 0 |  | 0
  Varicella: Swelling: Any Grade: number analyzed (Participants) | 103 | 0 | 53 | 86 | 0 | 42
  Varicella: Swelling: Any Grade | 10 |  | 2 | 12 |  | 5
  Varicella: Swelling: Grade 3: number analyzed (Participants) | 103 | 0 | 53 | 86 | 0 | 42
  Varicella: Swelling: Grade 3 | 0 |  | 0 | 0 |  | 0

14. Secondary Outcome: Number of Participants Reporting at Least One Solicited Injection Site Reactions (Tenderness, Erythema, and Swelling): Groups 4, 5, and 6
Description: SR was defined as an AE that was prelisted (i.e., solicited) in the eCRF and considered to be related to vaccination (adverse drug reaction). Solicited injection site reactions: tenderness, erythema, and swelling. Tenderness: Grade 3: cries when injected limb moved or the movement of the injected limb reduced, Erythema and swelling: Grade 3: >= 50 mm. Participants with any of the Grade and Grade 3 solicited injection-site reactions were reported.
Time Frame: Within 7 days post vaccination
Population: Analysis was performed on SafAS. Here, 'Number analyzed' = participants with available data for each specified category and '0' in the number analyzed field signifies that the vaccines mentioned in the respective categories were not administered to the specified group.
Measure: Count of Participants; unit: Participants
Arm/Group | Mexico (Group 4): MenACYW Conjugate + DTaP-IPV-HB-Hib Vaccine | Mexico (Group 5): MenACYW Conjugate Vaccine | Mexico (Group 6): DTaP-IPV-HB-Hib Vaccine
Number analyzed (Participants) | 200 | 100 | 100
Participants
  MenACYW: Tenderness: Any Grade: number analyzed (Participants) | 191 | 98 | 0
  MenACYW: Tenderness: Any Grade | 68 | 27 |
  MenACYW: Tenderness: Grade 3: number analyzed (Participants) | 191 | 98 | 0
  MenACYW: Tenderness: Grade 3 | 6 | 1 |
  MenACYW: Erythema: Any Grade: number analyzed (Participants) | 191 | 98 | 0
  MenACYW: Erythema: Any Grade | 40 | 15 |
  MenACYW: Erythema: Grade 3: number analyzed (Participants) | 191 | 98 | 0
  MenACYW: Erythema: Grade 3 | 3 | 3 |
  MenACYW: Swelling: Any Grade: number analyzed (Participants) | 191 | 98 | 0
  MenACYW: Swelling: Any Grade | 23 | 8 |
  MenACYW: Swelling: Grade 3: number analyzed (Participants) | 191 | 98 | 0
  MenACYW: Swelling: Grade 3 | 2 | 2 |
  DTaP-IPV-HB-Hib: Tenderness: Any Grade: number analyzed (Participants) | 191 | 0 | 95
  DTaP-IPV-HB-Hib: Tenderness: Any Grade | 80 |  | 54
  DTaP-IPV-HB-Hib: Tenderness: Grade 3: number analyzed (Participants) | 191 | 0 | 95
  DTaP-IPV-HB-Hib: Tenderness: Grade 3 | 6 |  | 10
  DTaP-IPV-HB-Hib: Erythema: Any Grade: number analyzed (Participants) | 191 | 0 | 95
  DTaP-IPV-HB-Hib: Erythema: Any Grade | 56 |  | 37
  DTaP-IPV-HB-Hib: Erythema: Grade 3: number analyzed (Participants) | 191 | 0 | 95
  DTaP-IPV-HB-Hib: Erythema: Grade 3 | 8 |  | 5
  DTaP-IPV-HB-Hib: Swelling: Any Grade: number analyzed (Participants) | 191 | 0 | 95
  DTaP-IPV-HB-Hib: Swelling: Any Grade | 45 |  | 30
  DTaP-IPV-HB-Hib: Swelling: Grade 3: number analyzed (Participants) | 191 | 0 | 95
  DTaP-IPV-HB-Hib: Swelling: Grade 3 | 8 |  | 4

15. Secondary Outcome: Number of Participants Reporting at Least One Solicited Injection Site Reactions (Tenderness, Erythema, and Swelling): Groups 7, 8, and 9
Description: SR was defined as an AE that was prelisted (i.e., solicited) in the eCRF and considered to be related to vaccination (adverse drug reaction). Solicited injection site reactions: tenderness, erythema, and swelling. Tenderness: Grade 3: cries when injected limb moved, or the movement of the injected limb reduced, Erythema and swelling: Grade 3: >= 50 mm. Participants with any of the Grade and Grade 3 solicited injection-site reactions were reported.
Time Frame: Within 7 days post vaccination
Population: Analysis was performed on SafAS. Here, '0' in the number analyzed field signifies that the vaccines mentioned in the respective categories were not administered to the specified group.
Measure: Count of Participants; unit: Participants
Arm/Group | Russian Federation (Group 7):MenACYW Conjugate + PCV13 Vaccine | Russian Federation (Group 8): MenACYW Conjugate Vaccine | Russian Federation (Group 9): PCV13 Vaccine
Number analyzed (Participants) | 200 | 100 | 99
Participants
  MenACYW: Tenderness: Any Grade: number analyzed (Participants) | 200 | 100 | 0
  MenACYW: Tenderness: Any Grade | 28 | 8 |
  MenACYW: Tenderness: Grade 3: number analyzed (Participants) | 200 | 100 | 0
  MenACYW: Tenderness: Grade 3 | 4 | 0 |
  MenACYW: Erythema: Any Grade: number analyzed (Participants) | 200 | 100 | 0
  MenACYW: Erythema: Any Grade | 43 | 17 |
  MenACYW: Erythema: Grade 3: number analyzed (Participants) | 200 | 100 | 0
  MenACYW: Erythema: Grade 3 | 0 | 0 |
  MenACYW: Swelling: Any Grade: number analyzed (Participants) | 200 | 100 | 0
  MenACYW: Swelling: Any Grade | 8 | 7 |
  MenACYW: Swelling: Grade 3: number analyzed (Participants) | 200 | 100 | 0
  MenACYW: Swelling: Grade 3 | 0 | 0 |
  PCV13: Tenderness: Any Grade: number analyzed (Participants) | 200 | 0 | 99
  PCV13: Tenderness: Any Grade | 34 |  | 9
  PCV13: Tenderness: Grade 3: number analyzed (Participants) | 200 | 0 | 99
  PCV13: Tenderness: Grade 3 | 5 |  | 1
  PCV13: Erythema: Any Grade: number analyzed (Participants) | 200 | 0 | 99
  PCV13: Erythema: Any Grade | 48 |  | 8
  PCV13: Erythema: Grade 3: number analyzed (Participants) | 200 | 0 | 99
  PCV13: Erythema: Grade 3 | 0 |  | 0
  PCV13: Swelling: Any Grade: number analyzed (Participants) | 200 | 0 | 99
  PCV13: Swelling: Any Grade | 19 |  | 2
  PCV13: Swelling: Grade 3: number analyzed (Participants) | 200 | 0 | 99
  PCV13: Swelling: Grade 3 | 0 |  | 0

16. Secondary Outcome: Number of Participants Reporting at Least One Solicited Systemic Reactions (Fever, Vomiting, Abnormal Crying, Drowsiness, Appetite Loss, and Irritability)
Description: SR was defined as an AE that was prelisted (i.e., solicited) in the eCRF and considered to be related to vaccination (adverse drug reaction). Solicited systemic reaction: Fever: Grade 3: > 39.5 degree Celsius, Vomiting: Grade 3: >= 6 episodes per 24 hours or requiring parenteral hydration, Crying abnormal: Grade 3: > 3 hours, Drowsiness: Grade 3: sleeping most of the time or difficult to wake up, Appetite lost: Grade 3: refuses >= 3 feeds/meals or refuses most feeds/meals, Irritability: Grade 3: inconsolable. Participants with any of the Grade and Grade 3 solicited systemic reactions were reported.
Time Frame: Within 7 days post vaccination
Population: Analysis was performed on Safety analysis set. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Russian Federation (Group7): MenACYW Conjugate + PCV13 Vaccine: Healthy, meningococcal-vaccine naïve toddlers (aged 15 to 23 months) received single dose of MenACYW Conjugate vaccine and PCV13 vaccine on Day 0.
Arm/Group | South Korea(Group1):MenACYW Conjugate +MMR +Varicella Vaccine | South Korea (Group 2): MenACYW Conjugate Vaccine | South Korea (Group 3): MMR + Varicella Vaccine | Thailand (Group 10):MenACYW Conjugate + MMR +Varicella Vaccine | Thailand (Group 11): MenACYW Conjugate Vaccine | Thailand (Group 12): MMR + Varicella Vaccine | Mexico (Group 4): MenACYW Conjugate + DTaP-IPV-HB-Hib Vaccine | Mexico (Group 5): MenACYW Conjugate Vaccine | Mexico (Group 6): DTaP-IPV-HB-Hib Vaccine | Russian Federation (Group7): MenACYW Conjugate + PCV13 Vaccine | Russian Federation (Group 8): MenACYW Conjugate Vaccine | Russian Federation (Group 9): PCV13 Vaccine
Number analyzed (Participants) | 103 | 52 | 53 | 86 | 42 | 42 | 191 | 98 | 95 | 200 | 100 | 99
Participants
  Fever: Any Grade | 17 | 9 | 5 | 6 | 1 | 3 | 32 | 7 | 16 | 12 | 3 | 2
  Fever: Grade 3 | 1 | 2 | 1 | 0 | 1 | 0 | 4 | 1 | 0 | 0 | 0 | 0
  Vomiting: Any Grade | 6 | 3 | 2 | 5 | 4 | 5 | 15 | 6 | 9 | 0 | 0 | 0
  Vomiting: Grade 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Abnormal crying: Any Grade | 21 | 9 | 6 | 14 | 17 | 12 | 46 | 25 | 26 | 8 | 4 | 2
  Abnormal crying: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 0
  Drowsiness: Any Grade | 17 | 8 | 9 | 8 | 7 | 7 | 31 | 15 | 17 | 25 | 6 | 4
  Drowsiness: Grade 3 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 0
  Appetite Lost: Any Grade | 29 | 10 | 8 | 11 | 12 | 5 | 51 | 25 | 20 | 19 | 12 | 7
  Appetite Lost: Grade 3 | 1 | 0 | 0 | 0 | 0 | 2 | 8 | 2 | 3 | 1 | 0 | 0
  Irritability: Any Grade | 31 | 12 | 11 | 14 | 11 | 14 | 64 | 34 | 33 | 26 | 16 | 9
  Irritability: Grade 3 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 1 | 3 | 4 | 0 | 0

ADVERSE EVENTS:
Time Frame: AE data were collected from Day 0 up to Day 30 post-vaccination. SR data were collected within 7 days after vaccination. Serious adverse event (SAE) data were collected throughout the study period (up to Day 30 post-vaccination).
Description: SR: an AE that was prelisted (i.e., solicited) in the eCRF and considered to be related to vaccination (adverse drug reaction). An unsolicited AE was an observed AE that did not fulfill the conditions prelisted in the eCRF (i.e., solicited) in terms of symptom and/or onset post-vaccination. Analysis was done on SafAS. In the AE section, solicited reactions Fever, Abnormal crying, Drowsiness, and Appetite lost are reported under Pyrexia, Crying, Somnolence, and Decreased Appetite, respectively.
Groups:
- South Korea(Group1):MenACYW Conjugate +MMR +Varicella Vaccine; Thailand (Group 10):MenACYW Conjugate + MMR +Varicella Vaccine: Healthy, meningococcal-vaccine naïve toddlers (aged 12 to 23 months) received single dose of MenACYW Conjugate vaccine, MMR vaccine, and varicella vaccine on Day 0.
- Russian Federation (Group 7):MenACYW Conjugate + PCV13 Vaccine: Healthy, meningococcal-vaccine naïve toddlers (aged 15 to 23 months) received single dose of MenACYW Conjugate and PCV13 Vaccine on Day 0.
Arm/Group | South Korea(Group1):MenACYW Conjugate +MMR +Varicella Vaccine | South Korea (Group 2): MenACYW Conjugate Vaccine | South Korea (Group 3): MMR + Varicella Vaccine | Thailand (Group 10):MenACYW Conjugate + MMR +Varicella Vaccine | Thailand (Group 11): MenACYW Conjugate Vaccine | Thailand (Group 12): MMR + Varicella Vaccine | Mexico (Group 4): MenACYW Conjugate + DTaP-IPV-HB-Hib Vaccine | Mexico (Group 5): MenACYW Conjugate Vaccine | Mexico (Group 6): DTaP-IPV-HB-Hib Vaccine | Russian Federation (Group 7):MenACYW Conjugate + PCV13 Vaccine | Russian Federation (Group 8): MenACYW Conjugate Vaccine | Russian Federation (Group 9): PCV13 Vaccine
All-Cause Mortality (participants affected / at risk) | 0/103 | 0/52 | 0/53 | 0/86 | 0/42 | 0/42 | 0/200 | 0/100 | 0/100 | 0/200 | 0/100 | 0/99
Serious Adverse Events (participants affected / at risk) | 6/103 | 4/52 | 2/53 | 0/86 | 1/42 | 0/42 | 0/200 | 0/100 | 1/100 | 0/200 | 0/100 | 0/99
Other Adverse Events (participants affected / at risk) | 85/103 | 43/52 | 37/53 | 58/86 | 37/42 | 37/42 | 142/200 | 65/100 | 85/100 | 75/200 | 30/100 | 17/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | South Korea(Group1):MenACYW Conjugate +MMR +Varicella Vaccine (N=103) | South Korea (Group 2): MenACYW Conjugate Vaccine (N=52) | South Korea (Group 3): MMR + Varicella Vaccine (N=53) | Thailand (Group 10):MenACYW Conjugate + MMR +Varicella Vaccine (N=86) | Thailand (Group 11): MenACYW Conjugate Vaccine (N=42) | Thailand (Group 12): MMR + Varicella Vaccine (N=42) | Mexico (Group 4): MenACYW Conjugate + DTaP-IPV-HB-Hib Vaccine (N=200) | Mexico (Group 5): MenACYW Conjugate Vaccine (N=100) | Mexico (Group 6): DTaP-IPV-HB-Hib Vaccine (N=100) | Russian Federation (Group 7):MenACYW Conjugate + PCV13 Vaccine (N=200) | Russian Federation (Group 8): MenACYW Conjugate Vaccine (N=100) | Russian Federation (Group 9): PCV13 Vaccine (N=99)
Bronchiolitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis Viral (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Croup Infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand-Foot-And-Mouth Disease (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis Media Viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia Viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory Syncytial Virus Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | South Korea(Group1):MenACYW Conjugate +MMR +Varicella Vaccine (N=103) | South Korea (Group 2): MenACYW Conjugate Vaccine (N=52) | South Korea (Group 3): MMR + Varicella Vaccine (N=53) | Thailand (Group 10):MenACYW Conjugate + MMR +Varicella Vaccine (N=86) | Thailand (Group 11): MenACYW Conjugate Vaccine (N=42) | Thailand (Group 12): MMR + Varicella Vaccine (N=42) | Mexico (Group 4): MenACYW Conjugate + DTaP-IPV-HB-Hib Vaccine (N=200) | Mexico (Group 5): MenACYW Conjugate Vaccine (N=100) | Mexico (Group 6): DTaP-IPV-HB-Hib Vaccine (N=100) | Russian Federation (Group 7):MenACYW Conjugate + PCV13 Vaccine (N=200) | Russian Federation (Group 8): MenACYW Conjugate Vaccine (N=100) | Russian Federation (Group 9): PCV13 Vaccine (N=99)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 12 (13) | 5 (6) | 6 (6) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 7 (7) | 3 (3) | 2 (2) | 6 (6) | 4 (4) | 6 (6) | 16 (17) | 7 (7) | 9 (9) | 0 (0) | 0 (0) | 0 (0) — Vomiting events that occurred after 7 days post-vaccination were considered as unsolicited AE.
Crying (General disorders) | 21 (21) | 9 (9) | 6 (6) | 15 (15) | 17 (17) | 12 (12) | 46 (46) | 25 (25) | 26 (26) | 8 (8) | 4 (4) | 2 (2) — Crying/Abnormal crying events that occurred after 7 days post-vaccination were considered as unsolicited AE.
Injection Site Erythema (General disorders) | 35 (60) | 20 (20) | 8 (10) | 36 (71) | 13 (13) | 16 (23) | 67 (96) | 15 (15) | 37 (37) | 55 (91) | 17 (17) | 8 (8)
Injection Site Pain (General disorders) | 31 (72) | 15 (15) | 12 (21) | 31 (63) | 17 (17) | 19 (32) | 87 (148) | 27 (27) | 54 (54) | 37 (62) | 8 (8) | 9 (9)
Injection Site Swelling (General disorders) | 25 (35) | 14 (14) | 3 (3) | 18 (38) | 7 (7) | 5 (9) | 52 (68) | 8 (8) | 30 (30) | 21 (27) | 7 (7) | 2 (2)
Pyrexia (General disorders) | 21 (21) | 11 (12) | 10 (12) | 6 (6) | 3 (3) | 4 (4) | 35 (35) | 8 (8) | 17 (17) | 13 (13) | 3 (3) | 2 (3) — Pyrexia/Fever events that occurred after 7 days post-vaccination were considered as unsolicited AE.
Bronchitis (Infections and infestations) | 4 (4) | 1 (1) | 4 (5) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 29 (37) | 17 (23) | 13 (18) | 5 (5) | 3 (4) | 6 (7) | 29 (31) | 18 (18) | 15 (16) | 2 (2) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 3 (4) | 2 (2) | 1 (1) | 2 (2) | 9 (9) | 6 (6) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 6 (6) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 6 (7) | 3 (3) | 0 (0) | 3 (3) | 2 (2) | 4 (4) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 29 (29) | 10 (10) | 8 (8) | 11 (11) | 12 (12) | 5 (5) | 51 (51) | 25 (25) | 20 (20) | 19 (19) | 12 (12) | 7 (7)
Somnolence (Nervous system disorders) | 17 (17) | 8 (8) | 9 (9) | 8 (8) | 7 (7) | 7 (7) | 31 (31) | 15 (15) | 17 (17) | 25 (25) | 6 (6) | 4 (4)
Irritability (Psychiatric disorders) | 31 (31) | 12 (12) | 11 (11) | 14 (15) | 11 (11) | 14 (14) | 64 (64) | 34 (34) | 33 (33) | 26 (26) | 16 (16) | 9 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2017-09-11): https://cdn.clinicaltrials.gov/large-docs/71/NCT03205371/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-29): https://cdn.clinicaltrials.gov/large-docs/71/NCT03205371/SAP_001.pdf